CLINICAL TRIAL: NCT00342940
Title: A Phase II, Open-Label, Uncontrolled, Single Center Study to Evaluate Safety and Immunogenicity of a Commercially Available Surface Antigen, Inactivated Influenza Vaccine, Formulation 2006-2007, When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Commercially Available Influenza Vaccine (Formulation 2006/2007) When Administered to Subjects 18 Years of Age or Older
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Vaccine Supplies
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V78P4S; Eudract number:2006-000787-88
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: influenza; influenza vaccine; flu; vaccination; immunogenicity
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: influenza surface antigen inactivated vaccine

SUMMARY:
The present study aims to evaluate safety and immunogenicity of one dose of a commercially available Surface Antigen, Inactivated Influenza Vaccine, Formulation 2006-2007, in non-elderly adult and elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 years of age or older

Exclusion Criteria:

* any auto-immune disease or other serious acute, chronic or progressive disease
* hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine
* known or suspected (or high risk of developing) impairment/alteration of immune function
* within the past 7 days any acute disease or infections requiring systemic antibiotic or antiviral therapy
* history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
CHMP criteria for evaluation of flu vaccines e.g Seroprotection, GMR's and Seroconversion rate at day 21 following vaccination

SECONDARY OUTCOMES:
Number and percentage of subjects with at least one local reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one systemic reaction between Day 0 and Day 3 after vaccine injection.
Number and percentage of subjects with at least one adverse event between Day 0 and the study termination visit (Day 21, window: 20-24).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines Drug Information Services, Study Chair — Novartis
Locations (1):
- Chiltern International Limited , Chiltern Place, Upton Road, Slough, United Kingdom